CLINICAL TRIAL: NCT04797741
Title: Adapting Internet Delivery of Enhanced Assess, Acknowledge, Act (IDEA3), an Evidence-based Sexual Assault Prevention Intervention for Women Undergraduates
Brief Title: Adapting an Evidence-based Sexual Assault Prevention Intervention for Women Undergraduates for Online Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sarah Melissa Peitzmeier, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00183965; 0920-1301 (Other Grant/Funding Number: National Center for Injury Prevention and Control)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Sexual Assault

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IDEA3 Intervention (Experimental)
  Interventions: Other: IDEA3 Intervention

INTERVENTIONS:
Other: IDEA3 Intervention — Delivery of IDEA3 intervention, a 12-hour online sexual assault resistance intervention for college women.

SUMMARY:
Sexual assault on college campuses is a prevalent public health problem, with 1 in 3 women experiencing sexual assault during her time in college. It is a major cause of injury, mental health concerns, sexually transmitted infections, and poor educational outcomes in youth and young adults. The Enhanced Assess, Acknowledge, Act (EAAA) sexual assault resistance intervention is the only intervention that has been shown to reduce sexual assault victimization for college women in a randomized controlled trial. EAAA is a 12-hour, peer facilitator-led, in-person intervention proven to reduce attempted or completed rape victimization by over 50% among female undergraduates, with durable effects lasting more than two years. Despite its unique efficacy, uptake of EAAA has been limited, in large part because universities prefer less costly interventions that can be administered online; unfortunately, no online intervention has been proven to reduce victimization.

This project seeks to adapt the existing EAAA intervention for online delivery to groups of students by live facilitators using a systematic adaptation process called ADAPT-ITT. After adapting and refining the intervention, the proposed work seeks to collect feasibility, acceptability, and efficacy-related outcome data.

The project has three aims:

1. Aim 1: Following the ADAPT-ITT framework, pilot a minimally adapted internet-delivered EAAA (IDEA3) with undergraduate women (n=12), collecting data on acceptability immediately following the intervention.
2. Aim 2: Produce a fully adapted IDEA3 intervention that retains core elements of the in-person intervention crucial for efficacy, while capitalizing on unique strengths of the online modality.
3. Aim 3: Test the feasibility and acceptability of IDEA3 through a pilot trial and examine intermediary outcomes shown to be strong mediators of EAAA's effect on reducing victimization (n=64).

The investigators hope this intervention may prevent as many as 50% of sexual assaults experienced by college women, comparable to the existing in-person intervention from which this online intervention is being adapted. Once the intervention has been finalized, the investigators plan to disseminate the intervention and make it widely available to institutions through the SARE Centre, a non-profit partner on the study that currently disseminates the in-person version of the intervention, EAAA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults ages 18 to 24, AND
* Identify as a woman, AND
* Be a first-year or second-year undergraduate student at the University of Michigan - Ann Arbor, AND
* Reside in Ann Arbor during the program, AND
* Be available during the program times, AND
* Provide the contact information for another woman undergraduate who they would be willing to participate in the intervention with OR express willingness to being partnered with another woman undergraduate at their university AND
* Have access to and willingness to use the videoconferencing software Zoom for the program AND
* Consent to being observed while participating.

Exclusion Criteria:

* Participant is less than 18 years of age or older than 24 years of age, OR
* Does not identify as a woman, OR
* Is not a first-year or second-year undergraduate student at the University of Michigan Ann Arbor, OR
* Does not reside in Ann Arbor, MI during the program, OR
* Is not available during the program times, OR
* Does not provide the contact information for another woman undergraduate who they would be willing to participate in the intervention with AND does not express a willingness to being partnered with another undergraduate OR
* Does not have access to and or is unwilling to use the videoconferencing software Zoom, OR
* Does not consent to being observed while participating.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is designed specifically for undergraduates who identify as women.
Enrollment: 76 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of IDEA3 intervention | Within one week of the final intervention session
  This will be assessed by reviewing speed of recruitment and noting no-shows (at first session), overall session attendance, and retention rates for the online intervention to determine whether incentives are sufficient for a future larger trial; reviewing fidelity to the original intervention based on reviewing recordings of all online intervention sessions; reviewing and cataloging deviations from the manual; and final review of what pieces of IDEA3 went well and what pieces need to be further adapted in the future.
Acceptability of IDEA3 intervention | Within one week of the final intervention session
  This will be assessed from summary statistics calculated from survey questions completed by participants relating to dimensions of affective attitude (how the individual feels about the intervention); burden (perceived effort required to participate); ethicality (extent to which the intervention fits with the individual's value system), perceived effectiveness, and whether they would recommend the intervention to a friend.
Intervention participants' self-defense self-efficacy | Within one week of the final intervention session
  This will be assessed from participant answers to baseline and post-test surveys that use validated scales to measure self-defense self-efficacy (i.e. confidence that one could defend oneself against sexual assault)

SECONDARY OUTCOMES:
Efficacy of IDEA3 intervention | Within one week of the final intervention session
  This will be assessed from participant answers to baseline and post-test surveys that use validated scales to measure five intermediary outcomes that account for EAAA's effect on reducing victimization: earlier detection of risk in coercive situations; greater risk perception of acquaintance rape; lower rape myth acceptance; knowledge of, and willingness to use evidence-based forceful verbal and physical resistance in a hypothetical situation; and earlier identification of 'discomfort' and earlier willingness to leave a hypothetical situation.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Peitzmeier, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data from video recordings contain identifiers including participant images and names which cannot be removed, and will therefore remain non-public. Deidentified survey data from initial screener surveys can be made available upon request.